CLINICAL TRIAL: NCT03562195
Title: A Randomized, Double Blind, Parallel Group Study of the Efficacy and Safety of Mepolizumab as Adjunctive Therapy in Patients With Severe Asthma With Eosinophilic Inflammation
Brief Title: A Safety and Efficacy Study of Mepolizumab in Subjects With Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201536
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: Eosinophilic inflammation; Mepolizumab; Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized in 1:1 ratio to receive either mepolizumab or placebo along with existing standard of care therapy during the treatment period.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mepolizumab 100mg (Experimental): Participants received 100mg of Mepolizumab subcutaneously every 4 weeks during the total treatment period of 52 weeks in addition to their baseline Standard of Care (SOC) treatment for asthma. Participants received salbutamol as a rescue medication on need basis.
  Interventions: Drug: Mepolizumab 100 milligrams; Drug: Salbutamol
- Placebo (Placebo Comparator): Participants received placebo matching to Mepolizumab administered subcutaneously every 4 weeks during the total treatment period of 52 weeks in addition to their baseline SOC treatment for asthma. Participants received salbutamol as a rescue medication on need basis
  Interventions: Drug: Placebo; Drug: Salbutamol

INTERVENTIONS:
Drug: Mepolizumab 100 milligrams — Mepolizumab will be given as a lyophilized cake in sterile vials for individual use. The vial will be reconstituted with Sterile Water for Injection, just prior to use.
  Arms: Mepolizumab 100mg
Drug: Placebo — Placebo will be given as 0.9 percent sodium chloride solution.
  Arms: Placebo
Drug: Salbutamol — Salbutamol MDI will be given as a rescue medication to be used on an as needed basis in this study.

SUMMARY:
Mepolizumab, a humanized monoclonal antibody, has been developed as an add-on treatment for subjects with severe asthma with eosinophilic inflammation. Current asthma treatment guidelines offer minimal options for the severe asthmatic subjects on intensive therapy with frequent exacerbations. There is a significant unmet medical need to provide better treatment options for this segment of the asthma population. Thus, this study is designed to evaluate the efficacy and safety of mepolizumab in Chinese severe asthmatic subjects with eosinophilic inflammation. A total number of 300 subjects will be randomized in 1:1 ratio to receive either mepolizumab or placebo along with existing standard of care therapy. The maximum study duration will be 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will be able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Subjects with at least 12 years of age at Visit 0 and a minimum weight of 40 kilograms.
* Persistent airflow obstruction as indicated by: For subjects >=18 years of age at visit 1, a pre-bronchodilator FEV1 <80 percent predicted (National Health and Nutrition Examination Survey [NHANES] III).;For subjects 12 to 17 years of age at Visit 1: A pre-bronchodilator FEV1 <90 percent predicted (NHANES III) recorded at Visit 1 or FEV1: Forced vital capacity (FVC) ratio <0.8 recorded at Visit 1.
* Prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma as per Randomization Criteria 1 (Documented peripheral blood eosinophil count of >=300 cells per microliters that is related to asthma in the past 12 months prior to Visit 1 or a peripheral blood eosinophil count of >=150 cells per microliters at Visit 1 that is related to asthma).
* Regular treatment with high dose inhaled corticosteroid (ICS) in the 12 months prior to Visit 1, of which at least 9 months accumulated documented is required, the 3 months prior to Visit 1 is mandatory. With or without maintenance oral corticosteroids (OCS). ICS dose must be >=500 microgram per day fluticasone propionate (FP) or equivalent daily (for ICS/long-acting beta-2-agonists combination preparations, Seretide 50/250 micrograms twice daily and above or equivalent will meet this ICS criteria). (Maintenance OCS is defined as a prescribed regimen of a minimum average daily dose of prednisone 5 milligrams [or equivalent]).
* Current treatment with an additional controller medication, besides ICS, for at least 3 months. (Example given [e.g.], long-acting beta-2-agonist, leukotriene receptor antagonist [LTRA], or theophylline).
* Previously confirmed history of two or more exacerbations requiring treatment with systemic corticosteroid (intramuscular [IM], intravenous, or oral), in the 12 months prior to Visit 1, despite the use of high-dose ICS. For subjects receiving maintenance corticosteroid, the corticosteroid treatment for the exacerbations must have been a two-fold increase or greater in the dose for at least 3 days is required.
* A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1 percent, during the intervention period and for at least 4 months after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

A WOCBP must have a negative highly sensitive pregnancy test before the first dose of study intervention. If urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the subject must be excluded from participation if the serum pregnancy result is positive. Follicle-stimulating hormone will be assessed to confirm child-bearing status as needed in non WOCBP.

Exclusion Criteria:

* Current smokers or former smokers with a smoking history of >=10 pack years (number of pack years = (number of cigarettes per day/20) x number of years smoked). A former smoker is defined as a subject who quit smoking at least 6 months prior to Visit 1.
* Presence of a known pre-existing, clinically significant lung condition other than asthma, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study. This includes current bacterial or viral infection of the upper or lower respiratory tract, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer. Clinically Significant is defined as any disease/condition that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* A chest X-ray that reveals evidence of clinically significant abnormalities not believed to be due to the presence of asthma.
* Bronchial Thermoplasty and Radiotherapy are excluded for 12 months prior to visit 1 and throughout the study.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (Subjects that had localized carcinoma of the skin which was resected for cure will not be excluded).
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice or cirrhosis. Subjects with ALT >2 times Upper Limit of Normal (ULN), bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent)
* Subjects who have known, pre-existing severe or clinically significant cardiovascular disease uncontrolled with standard treatment. Including but not limited to: known ejection fraction of <30 percent or severe heart failure meeting New York Heart Association Class IV classification or hospitalized in the 12 months prior to Visit 1 for severe heart failure meeting New York Heart Association Class III or angina diagnosed less than 3 months prior to Visit 1 or at Visit 1.
* QT interval corrected by Fridericia's formula (QTc[F]) >450 milliseconds (msec) or QTc(F) >480 msec for subjects with Bundle Branch Block at Visit 1 is exclusive.
* Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, hematological or any other system abnormalities that are uncontrolled with standard treatment. Current malignancy except for basal and squamous skin cancer.
* Subjects with other conditions that could lead to elevated eosinophils such as Hypereosiniophilic Syndromes, including Churg-Strauss Syndrome, or Eosinophilic Esophagitis.
* Subjects with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 are also excluded.
* A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1. Alcohol abuse is defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than three units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than two units (females). One unit was equivalent to a half-pint (220 milliliters) of beer or one (25 milliliters) measure of spirits or one glass (125 milliliters) of wine.
* A known immunodeficiency (e.g., human immunodeficiency virus - HIV), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Subjects who have received omalizumab (Xolair) within 130 days of Visit 1.
* Subjects who have received any monoclonal antibodies (other than Xolair) to treat inflammatory disease within 5 half-lives of Visit 1.
* Use of herbals within 7 days prior to visit 1, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subjects who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to visit 1 (this also includes investigational formulations of marketed products).
* Subjects with allergy/intolerance to a monoclonal antibody or biologic.
* Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* Previously participated in any study with mepolizumab and received investigational product (including placebo).
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study. Re-screening of subjects will be allowed only upon approval by the medical monitor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- China (29):
  - GSK Investigational Site, Fuzhou, Fujian
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Guiyang, Guizhou
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Zhengzhou, Henan
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Hengyang, Hunan
  - GSK Investigational Site, Hohhot, Inner Mongolia
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Wuxi, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Ürümqi, Xinjiang
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Wenzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Chen R, Wei L, Dai Y, Wang Z, Yang D, Jin M, Xiong C, Li T, Hu S, Song J, Chan R, Kumar S, Abdelkarim A, Zhong N. Efficacy and safety of mepolizumab in a Chinese population with severe asthma: a phase III, randomised, double-blind, placebo-controlled trial. ERJ Open Res. 2024 May 20;10(3):00750-2023. doi: 10.1183/23120541.00750-2023. eCollection 2024 May. PMID 38770009
- [Derived] Chen R, Dai Y, Yang D, Liu C, Han W, Gu W, Cao J, Zhou Q, Howarth P, Weng S, Xiong C, Huang J, Liang P, Zhong N; 201536 Study Group. Clinical Remission Outcome in Chinese Patients With Severe Asthma With an Eosinophilic Phenotype Receiving Mepolizumab: A Post-hoc Analysis of a Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial. Allergy Asthma Immunol Res. 2025 Jul;17(4):473-485. doi: 10.4168/aair.2025.17.4.473. PMID 40736776

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 371 participants with severe asthma and eosinophilic inflammation who meet the protocol defined inclusion criteria were screened. Off these, 300 participants were randomized in 1:1 ratio to mepolizumab: placebo arms. 149 participants in the mepolizumab treatment group and 151 participants in the placebo treatment group.
Period: Overall Study
Arm/Group | Mepolizumab 100mg | Placebo
Started | 149 | 151
Completed | 145 | 138
Not Completed | 4 | 13
Not completed — Adverse Event | 0 | 6
Not completed — Lack of Efficacy | 0 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 100mg | Placebo | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (12.59) | 53.7 (13.59) | 52.2 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 83 | 164
  Male | 68 | 68 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 149 | 151 | 300

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinically Significant Exacerbations of Asthma
Description: Clinically significant exacerbation is defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalizations and/or Emergency Department (ED) visits. Analysis of the number of exacerbations was performed using a negative binomial model with covariates of treatment group, baseline maintenance Oral Corticosteroids (OCS) therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted Forced Expiratory Volume in 1 second (FEV1), and with logarithm of time on treatment as an offset variable.
Time Frame: Up to Week 52
Population: The analysis was performed on the Modified Intent-to-Treat (MITT) Set that included all randomized participants who received at least one dose of trial medication. 'Modified' implies that participants who were randomized but did not receive study treatment were excluded.
Measure: Number; unit: Exacerbations per year
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Exacerbations per year | 0.45 | 1.31
Statistical Analysis 1: Comparison: Mepolizumab 100mg vs Placebo; Test type: Superiority; Bayesian Dynamic Borrowing; A BDB approach was used in the estimation of primary endpoint in the Chinese participants of this study, with information borrowed from MEA115588; Posterior probablity = 0.9999 — Pr (rate ratio <1 | data)>0.999. The 'positive result' is defined as if the posterior probability that the rate ratio is less than 1 is at least 0.95
Statistical Analysis 2: Comparison: Mepolizumab 100mg vs Placebo; Test type: Superiority — The null hypothesis is defined as the rate ratio of events between Mepolizumab 100mg SC versus placebo is less than 1; p < 0.001, Negative binomial model; Rate Ratio = 0.35, 95% CI 2-sided [0.24 to 0.50]

2. Secondary Outcome: Percent Probability of First Clinically Significant Exacerbations at Week 16, Week 32, and Week 52
Description: Clinically significant exacerbation is defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalizations and/or Emergency Department (ED) visits. Analysis of the number of exacerbations was performed using a negative binomial model with covariates of treatment group, baseline maintenance Oral Corticosteroids (OCS) therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted Forced Expiratory Volume in 1 second (FEV1), and with logarithm of time on treatment as an offset variable. Time to first clinically significant exacerbation was analyzed using Kaplan-Meier estimates and expressed in terms of probability.
Time Frame: Week 16, 32 and 52
Population: The analysis was performed on the MITT Set that included all randomized participants who received at least one dose of trial medication. 'Modified' implies that participants who were randomized but did not receive study treatment were excluded.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Percent probability
  Week 16 | 14.1 [9.43 to 20.79] | 34.7 [27.64 to 42.87]
  Week 32 | 18.1 [12.82 to 25.32] | 47.9 [40.18 to 56.25]
  Week 52 | 28.4 [21.86 to 36.44] | 53.6 [45.74 to 61.84]

3. Secondary Outcome: Mean Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) at Week 52
Description: The SGRQ Questionnaire is a well-established, self-completed tool, with 50 questions comprising three domains: Symptoms, Activity, and Impacts scores (each ranging from 0 to 100; where higher score indicates worst outcome). SGRQ total score was calculated by summing weights from all positive items, divided by sum of weights for all items in SGRQ questionnaire and multiplying by 100. The SGRQ total score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Analysis was performed using mixed model repeated measures with covariates of baseline, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), baseline % predicted FEV1, treatment and visit, plus interaction terms for visit by baseline and visit by treatment group.
Time Frame: Baseline and Week 52
Population: The analysis was performed on the MITT Set that included all randomized participants who received at least one dose of trial medication. 'Modified' implies that participants who were randomized but did not receive study treatment were excluded. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 136 | 124
Scores on a scale | -14.29 (1.526) | -7.20 (1.577)

4. Secondary Outcome: Number of Participants With Clinically Significant Exacerbations Requiring Hospitalization (Including Intubation and Admittance to an Intensive Care Unit [ICU]) or Emergency Department (ED) Visits
Description: An exacerbation is defined as worsening of asthma requiring the use of systemic corticosteroids and/or emergency department visit, or hospitalization. The number of exacerbations requiring hospitalization including incubation and admittance to an Intensive care unit (ICU) or ED visits were evaluated. Analysis of number of exacerbations was performed using a negative binomial model with covariates of treatment group, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted FEV1, and with logarithm of time on treatment as an offset variable. The data for participants with 0, 1, 2 and 3 exacerbations requiring hospitalization (including intubation and admittance to an ICU) or ED visits are summarized.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Participants
  0 exacerbation | 144 | 133
  1 exacerbation | 3 | 14
  2 exacerbations | 2 | 3
  3 exacerbations | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant Exacerbations Requiring Hospitalization
Description: An exacerbation is defined as worsening of asthma requiring the use of systemic corticosteroids and/or emergency department visit, or hospitalization. Analysis of number of exacerbations was performed using a negative binomial model with covariates of treatment group, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted FEV1, and with logarithm of time on treatment as an offset variable. The summary data for participants with 0, 1, 2 and 3 exacerbations requiring hospitalization are summarized.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Participants
  0 exacerbation | 145 | 139
  1 exacerbation | 3 | 10
  2 exacerbations | 1 | 1
  3 exacerbations | 0 | 1

6. Secondary Outcome: Mean Change From Baseline in Clinic Prebronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 52
Description: FEV1 is the volume of air that can be forced out in one second after taking a deep breath. Prebronchodilator FEV1 were measured via spirometer at Baseline and Week 52. Analysis was performed using mixed model repeated measures with covariates of baseline, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), treatment and visit, plus interaction terms for visit by baseline and visit by treatment group.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Milliliter (mL)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 130 | 114
Milliliter (mL) | 262.79 (34.341) | 125.67 (35.488)

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) Including Systemic (i.e., Allergic [Type I Hypersensitivity] and Other Systemic) and Injection Site Reactions
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Systemic reactions and local injection site reactions are adverse events of special interest (AESIs).
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Participants
  Participants with AE | 135 | 146
  Participants with Systemic Reactions | 4 | 2
  Participants with Local Injection Site Reactions | 3 | 2

8. Secondary Outcome: Change From Baseline in Platelets Count
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter Platelets count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 127
Giga cells per liter (10^9/L) | 0.6 (35.46) | -3.5 (45.09)

9. Secondary Outcome: Change From Baseline in Erythrocytes Count
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter Erythrocytes count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tera cells per liter (10^12/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 127
Tera cells per liter (10^12/L) | -0.03 (0.257) | -0.05 (0.257)

10. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter Hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 127
Fraction of 1 | -0.004 (0.0257) | -0.003 (0.0260)

11. Secondary Outcome: Percent Change From Baseline in Mean White Blood Cell (WBC) Count With Differential (Neutrophils, Lymphocytes, Monocytes. Eosinophils and Basophils)
Description: Blood samples was collected for the assessment of change from baseline in WBC) count with differential (neutrophils, lymphocytes, monocytes. eosinophils and basophils). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Median (Full Range); unit: Percent change
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 127
Percent change
  Basophils/Leukocytes | 0.00 [-1.0 to 1.2] | 0.20 [-0.8 to 1.3]
  Eosinophils/Leukocytes | -4.95 [-26.4 to 5.3] | -0.80 [-13.8 to 15.1]
  Lymphocytes/Leukocytes | 0.45 [-20.8 to 17.3] | 0.20 [-26.4 to 15.1]
  Monocytes/Leukocytes | 0.30 [-5.4 to 4.3] | 0.30 [-16.7 to 5.9]
  Neutrophils/Leukocytes | 4.65 [-18.7 to 28.0] | -0.50 [-16.7 to 35.4]

12. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: Blood samples was collected for the assessment of change from baseline in clinical parameter Alkaline Phosphatase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Unit per Liter (IU/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 128
International Unit per Liter (IU/L) | 2.8 (16.16) | 1.5 (12.79)

13. Secondary Outcome: Change From Baseline in Alanine Aminotransferase and Aspartate Aminotransferase
Description: Blood samples was collected for the assessment of change from baseline in clinical parameter Alanine Aminotransferase, Aspartate Aminotransferase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 128
Units per liter (U/L)
  Alanine Aminotransferase | 0.8 (11.49) | 0.0 (10.77)
  Aspartate Aminotransferase | 1.5 (7.38) | -0.1 (6.31)

14. Secondary Outcome: Change From Baseline in Albumin and Total Protein
Description: Blood samples was collected for the assessment of change from baseline in clinical parameter albumin, total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 128
Gram per liter (g/L)
  Albumin | 0.1 (2.55) | -0.4 (2.39)
  Total Protein | -0.6 (3.53) | -0.6 (3.70)

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples was collected for the assessment of change from baseline in clinical parameter including total and direct bilirubin, creatinine, glucose, calcium, sodium, potassium, urea. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 52
Population: The analysis was performed on the MITT Set that included all randomized participants who received at least one dose of trial medication. 'Modified' implies that participants who were randomized but did not receive study treatment were excluded. Number of participants analyzed signifies those participants who were evaluable for this outcome measure. Here 'number analyzed' signifies those participants who were evaluated at specified category.
Measure: Mean (Standard Deviation); unit: Micro moles per liter (umol/L)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 142 | 128
Micro moles per liter (umol/L)
  Total Bilirubin | -0.1 (3.47) | -0.7 (3.43)
  Calcium | 0.014 (0.0874) | 0.016 (0.0773)
  Creatinine | -0.7 (6.89) | -0.9 (6.55)
  Direct Bilirubin: number analyzed (Participants) | 141 | 127
  Direct Bilirubin | 0.4 (0.55) | 0.3 (0.60)
  Glucose | 0.16 (0.921) | 0.09 (1.448)
  Potassium | 0.00 (0.350) | -0.04 (0.328)
  Sodium | -0.8 (2.42) | -0.7 (2.39)
  Urea | 0.205 (1.3284) | -0.058 (1.2335)

16. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in a sitting position after 5 minutes rest. The normal range for SBP is 90-140 mmHg and DBP is 60-90 millimeters of mercury (mmHg).
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 143 | 131
Millimeters of mercury (mmHg)
  Diastolic Blood Pressure, Week 52 | -0.9 (9.58) | -1.1 (8.42)
  Systolic Blood Pressure, Week 52 | -1.3 (12.46) | -0.5 (10.75)

17. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: Pulse rate measurement were measured in a sitting position after 5 minutes rest.
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 143 | 131
Beats per minute (bpm) | -1.3 (9.71) | -1.1 (10.14)

18. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: 12-Lead electrocardiogram (ECG) measurements were obtained after the participants had rested in the supine position for 5 minutes. Clinically significant abnormal findings are based on the judgement of the investigator.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 143 | 131
Participants | 7 | 13

19. Secondary Outcome: Number of Participants With Positive Anti-Mepolizumab Antibody
Description: Blood samples were collected for detection of binding and neutralizing anti-mepolizumab antibodies. Samples with a positive screening result continued for confirmation analysis. Samples with a positive confirmation analysis were considered positive for mepolizumab Anti-drug antibody (ADA).
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100mg | Placebo
Number analyzed (Participants) | 149 | 151
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: Serious adverse events (SAEs), Non-serious AEs and All-cause mortality were collected using modified Intent-to-Treat (MITT) population, comprised of all randomized participants who receive at least one dose of trial medication. 'Modified' implies that participants who were randomized but did not receive study treatment were excluded.
Arm/Group | Mepolizumab 100mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/149 | 2/151
Serious Adverse Events (participants affected / at risk) | 18/149 | 25/151
Other Adverse Events (participants affected / at risk) | 134/149 | 146/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100mg (N=149) | Placebo (N=151)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 5
Bronchitis (Infections and infestations) | 0 | 2
Chronic sinusitis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Central nervous system infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection 1 (<1%) 0 (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Sinusitis fungal (Infections and infestations) | 1 | 0
Cataract (Eye disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100mg (N=149) | Placebo (N=151)
Asthma (Respiratory, thoracic and mediastinal disorders) | 45 | 82
Upper respiratory tract infection (Infections and infestations) | 61 | 63
Nasopharyngitis (Infections and infestations) | 25 | 27
Bronchitis (Infections and infestations) | 17 | 14
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Headache (Nervous system disorders) | 8 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Dizziness (Nervous system disorders) | 11 | 6
Pharyngitis (Infections and infestations) | 10 | 7
Rhinitis (Infections and infestations) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Pneumonia (Infections and infestations) | 5 | 9
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 | 7
Pyrexia (General disorders) | 6 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3
Respiratory tract infection (Infections and infestations) | 3 | 7
Toothache (Gastrointestinal disorders) | 4 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 4
Conjunctivitis (Infections and infestations) | 2 | 6
Gastritis (Gastrointestinal disorders) | 3 | 5
Hypertension (Vascular disorders) | 2 | 6
Chronic gastritis (Gastrointestinal disorders) | 1 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 5
Otitis media (Infections and infestations) | 2 | 5
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Acute sinusitis (Infections and infestations) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03562195/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03562195/SAP_001.pdf